CLINICAL TRIAL: NCT03280225
Title: Risk Stratified Enhancements to Clinical Care: Targeting Care for Patients Identified Through Predictive Modeling as Being at High Risk for Suicide, With the Office of Mental Health Operations
Brief Title: REACH VET Implementation Program Evaluation
Acronym: REACH VET
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: SDR 16-195
Record Dates: First submitted 2017-09-06; First posted 2017-09-12 (Actual); Results first posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-05

CONDITIONS: Suicide
Keywords: Suicide; Prevention; Implementation; Facilitation
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: None Retained — No biospecimens will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- VAMC's receiving implementation support for REACH VET: This cohort consists of 28 VA Medical Centers (VAMC's) needing additional implementation support to fully implement REACH VET as identified by Veteran Integrated Service Network (VISN) leadership, and that agreed to participate.
  Interventions: Other: External facilitation

INTERVENTIONS:
Other: External facilitation — Facilitation is an evidence-based implementation strategy to support sites that have difficulty implementing innovative programs. Facilitation is a multi-faceted "process of interactive problem solving and support that occurs in the context of a recognized need for improvement and a supportive interpersonal relationship (Powell et al., 2015)." Facilitation has been used nationally across VA to implement a number of different clinical interventions. The current project will examine this minimally intensive version of implementation facilitation, virtual external facilitation.
  Other Names: Virtual external facilitation, facilitation, implementation facilitation

SUMMARY:
The VA's Office of Mental Health and Suicide Prevention implemented an new program to increase suicide prevention outreach for Veterans at highest risk for suicide. Using a statistical model, REACH VET, short for Recovery Engagement and Coordination for Health - Veterans Enhanced Treatment, uses information from Veterans' health records to identify those who are at a higher risk for suicide, hospitalization, illness, or other negative outcomes. Once a Veteran is identified, his or her VA mental health or primary care provider reaches out to check on the Veteran's well-being and review their treatment plan to determine if enhanced care is needed. The goal of the current study was to evaluate the implementation of this program. The objectives of this evaluation were to evaluate how well this program is put into place using an implementation strategy called virtual external facilitation, and to collect data about the cost of the program and the strategy.

DETAILED DESCRIPTION:
The VA's Office of Mental Health and Suicide Prevention is implemented an innovative new program to increase suicide prevention outreach and target Veterans at highest risk for suicide. Using a new predictive model, REACH VET, short for Recovery Engagement and Coordination for Health - Veterans Enhanced Treatment, analyzes existing data from Veterans' health records to identify those who are at a statistically elevated risk for suicide, hospitalization, illness, or other adverse outcomes. Once a Veteran is identified, their VA mental health or primary care provider reaches out to check on the Veteran's well-being and review their condition(s) and treatment plans to determine if enhanced care is needed.

The goal of the proposed study is to evaluate the implementation of REACH VET. The objectives of this evaluation are to:

1. evaluate the implementation of REACH VET using virtual external facilitation, and
2. collect preliminary data about the cost and cost offsets.

The current evaluation will examine the impact of a virtual external facilitation strategy on the implementation of REACH VET in 28 medical facilities across 7 Veteran Integrated Service Networks (VISNs) in a stepped wedge design. Primary implementation outcomes include metrics of REACH VET implementation: coordinator assignment, provider assignment, care evaluation, and attempted outreach. Qualitative interviews will be conducted with implementation facilitators, Suicide Prevention Coordinator(s), clinical leadership, and providers to identify barriers and facilitators to implementation of REACH VET and the experience of facilitation. Secondary data will be collected on the cost of the intervention and the cost of implementation strategy.

ELIGIBILITY:
Inclusion Criteria:

* VA employee at a facility receiving virtual external facilitation
* Involved in REACH VET implementation

Exclusion Criteria:

* Not a VA employee
* Not employed at a facility receiving virtual external facilitation
* Not involved in REACH VET implementation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include facilities receiving virtual external facilitation for REACH VET
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara J. Landes, PhD, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR
Locations (2):
- United States (2):
  - Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, North Little Rock, Arkansas
  - VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reger MA, Luxton DD, Tucker R, Comtois KA, Keen AD, Landes SJ, Matarazzo BB, Thompson C. Implementation Methods for the Caring Contacts Suicide Prevention Intervention. Professional Psychology, Research and Practice. 2017 Oct 1; 48(5):369-377.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: VA Medical Centers in five Veteran Integrated Service Networks were identified by leadership as needing additional support in or der to implement REACH VET.
Pre-assignment Details: This study focuses on the implementation of an innovative new program to increase suicide prevention within VHA. Twenty-eight (28) VHA medical facilities were identified by leadership from seven Veteran Integrated Service Networks (VISN) for implementation based upon need for additional support in standing up the program. All outcomes were reported at the facility level. No patients were enrolled in this study and no outcomes are reported at the patient level.
Units Other Than Participants: VAMC
Groups:
- VAMC's Receiving Implementation Support for REACH VET: 28 VA Medical Centers were chosen by leadership across seven VISN's for support implementing REACH VET.
  External facilitation: Facilitation is an evidence-based implementation strategy to support sites that have difficulty implementing innovative programs. Facilitation is a multi-faceted "process of interactive problem solving and support that occurs in the context of a recognized need for improvement and a supportive interpersonal relationship (Powell et al., 2015)." Facilitation has been used nationally across VA to implement a number of different clinical interventions. The current project will examine this minimally intensive version of implementation facilitation, virtual external facilitation.
Period: Overall Study
Arm/Group | VAMC's Receiving Implementation Support for REACH VET
Started | NA; 28 VAMC (Participants are not enrolled in this study. All enrollment and analysis were conducted at the VAMC level.)
Completed | NA; 23 VAMC (Five VAMC's began implementation of REACH VET prior to scheduled facilitation due to latency in scheduling and were thus dropped from the study. Study was conducted at the unit (VAMC) level, not participant level.)
Not Completed | NA; 5 VAMC

BASELINE CHARACTERISTICS:
Population: 23 VA Medical Centers participating in implementation of REACH VET, Participants were not assigned to study arms
Units Other Than Participants: VAMC
Groups:
- VISNs Requesting Implementation Support: This cohort consists of VA Medical Centers (VAMC's) needing additional implementation support to fully implement REACH VET as identified by Veteran Integrated Service Network (VISN) leadership, and that agreed to participate.
  External facilitation: Facilitation is an evidence-based implementation strategy to support sites that have difficulty implementing innovative programs. Facilitation is a multi-faceted "process of interactive problem solving and support that occurs in the context of a recognized need for improvement and a supportive interpersonal relationship (Powell et al., 2015)." Facilitation has been used nationally across VA to implement a number of different clinical interventions. The current project will examine this minimally intensive version of implementation facilitation, virtual external facilitation.
Arm/Group | VISNs Requesting Implementation Support
Number analyzed (Participants) | NA
Number analyzed (VAMC) | 23
Age, Continuous [Mean (Standard Deviation); unit: VAMC] | NA (NA) — Analysis was conducted at the facility level using aggregated data. Age was not collected from the aggregated data.
Sex: Female, Male [Count of Units; unit: VAMC]
  Female | NA — Analysis was conducted at the facility level using aggregated data. Sex was not collected from the aggregated data.
  Male | NA — Analysis was conducted at the facility level using aggregated data. Sex was not collected from the aggregated data.
Race/Ethnicity, Customized [Count of Units; unit: VAMC]
  Units | NA — Participants were not assigned to study arms
Coordinator Accepted Pre-Implementation [Mean (Standard Deviation); unit: percent] — The average percentage of eligible Veterans across all 23 participating sites having a coordinator assigned within 2 weeks of the monthly REACH VET report being released during the 6 month pre-implementation period.
  percent | 88.5 (16.7)
Provider Assigned Pre-Implementation [Mean (Standard Deviation); unit: percentage] — The average percentage of eligible Veterans across all 23 participating sites having a provider assigned within 2 weeks of the monthly REACH VET report being released during the 6 month pre-implementation period.
  percentage | 68.1 (25.5)
Care Evaluation Performed Pre-Implementation [Mean (Standard Deviation); unit: percentage] — The average percentage of eligible Veterans across all 23 participating sites receiving a care evaluation within 2 weeks of the monthly REACH VET report being released during the 6 month pre-implementation period.
  percentage | 63.4 (23.9)
Outreach Attempted Pre-Implementation [Mean (Standard Deviation); unit: percent] — The average percentage of eligible Veterans across all 23 participating sites where outreach was attempted within 2 weeks of the monthly REACH VET report being released during the 6 month pre-implementation period.
  percent | 56.2 (77.0)

OUTCOME MEASURES:

1. Primary Outcome: Coordinator Assigned Post-Implementation
Description: The average percentage of eligible Veterans across all 23 participating sites having a coordinator assigned within 2 weeks of the monthly REACH VET report being released during the 6 month post-implementation period.
Time Frame: 6 months after implementation was completed
Population: Data not collected at the participant level
Measure: Mean (Standard Deviation); unit: percentage
Units Other Than Participants: VAMC
Arm/Group | VISNs Requesting Implementation Support
Number analyzed (Participants) | NA
Number analyzed (VAMC) | 23
percentage | 97.6 (1.0)
Statistical Analysis 1: Comparison: VISNs Requesting Implementation Support; Odds Ratio of eligible Veterans being assigned a coordinator during the 6 month period following implementation compared to eligible Veterans being assigned a coordinator in the 6 month period prior to implementation; Test type: Other; p = .302, Regression, Logistic; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.73 to 2.82] — Odds ratios were estimated using GEE to control for clustering within VAMCs. Fixed effects included a time-dependent variable (pre-post) as well an independent variable of time to account for improvement due to secular trends

2. Primary Outcome: Provider Assigned Post-Implementation
Description: The average percentage of eligible Veterans across all 23 participating sites having a provider assigned within 2 weeks of the monthly REACH VET report being released during the 6 month post-implementation period .
Time Frame: 6 month period following implementation
Population: Data not collected at the participant level
Measure: Mean (Standard Deviation); unit: percent
Units Other Than Participants: VAMC
Arm/Group | VISNs Requesting Implementation Support
Number analyzed (Participants) | NA
Number analyzed (VAMC) | 23
percent | 87.2 (17.3)
Statistical Analysis 1: Comparison: VISNs Requesting Implementation Support; Odds Ratio of eligible Veterans being assigned a provider during the 6 month period following implementation compared to eligible Veterans being assigned a provider in the 6 month period prior to implementation; Test type: Other; p = 0.226, Regression, Logistic; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.86 to 1.93] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Care Evaluation Performed Post-Implementation
Description: The average percentage of eligible Veterans across all 23 participating sites receiving a care evaluation within 2 weeks of the monthly REACH VET report being released during the 6 month post-implementation period.
Time Frame: 6 month period following implementation
Population: Data not collected at the participant level
Measure: Mean (Standard Deviation); unit: percent
Units Other Than Participants: VAMC
Arm/Group | VISNs Requesting Implementation Support
Number analyzed (Participants) | NA
Number analyzed (VAMC) | 23
percent | 83.6 (18.9)
Statistical Analysis 1: Comparison: VISNs Requesting Implementation Support; Odds Ratio of eligible Veterans receiving a care evaluation during the 6 month period following implementation compared to eligible Veterans receiving a care evaluation in the 6 month period prior to implementation; Test type: Other; p = 0.199, Regression, Logistic; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.90 to 1.70] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Attempted Outreach Post-Implementation
Description: The average percentage of eligible Veterans across all 23 participating sites where outreach was attempted within 2 weeks of the monthly REACH VET report being released during the 6 month post-implementation period.
Time Frame: 6 month period following implementation
Population: Data not collected at the participant level
Measure: Mean (Standard Deviation); unit: percent
Units Other Than Participants: VAMC
Arm/Group | VISNs Requesting Implementation Support
Number analyzed (Participants) | NA
Number analyzed (VAMC) | 23
percent | 77.0 (20.6)
Statistical Analysis 1: Comparison: VISNs Requesting Implementation Support; Odds Ratio of eligible Veterans where outreach was attempted during the 6 month period following implementation compared to eligible Veterans where outreach was attempted in the 6 month period prior to implementation; Test type: Other; p = 0.011, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [1.08 to 1.76] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Organizational Readiness for Change Survey
Description: Eligible staff at participating VA facilities were solicited to complete a modified version of the Texas Christian University Organizational Readiness for Change - Staff (TCU ORC-S). We abbreviated the original instrument to 62 items and modified text for contextual relevance. Responses were collected from 22 sites across five Veteran Integrated Service Networks (VISN). The responses were scored on ten scales: Program Needs (10 - 50 higher is preferred), Training Needs (10 - 50 higher is preferred), Pressure for Change (10 - 50 higher is preferred), Staffing (10 - 50 higher is preferred), Mission (10 - 50 higher is preferred), Cohesion (10 - 50 higher is preferred), Autonomy (10 - 50 higher is preferred), Communication (10 - 50 higher is preferred), Stress (10 - 50 lower is preferred) and Change (10 - 50 lower is preferred).
Time Frame: 1 month
Population: Eligible staff from all participating facilities were solicited to complete the modified Texas Christian University Organizational Readiness for Change for Staff (TCU ORC-S). Eligible staff were not considered enrolled but did contribute to this assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: VAMC
Groups:
- VISN A: This VISN group consisted of 23 respondents from 4 of the 23 VAMCs.
- VISN B: This VISN group consisted of 55 respondents from 4 of the 23 VAMCs.
- VISN C: This VISN group consisted of 7 respondents from 2 of the 23 VAMCs with an additional 2 VAMC's in this VISN not responding.
- VISN D: This group consisted of 59 respondents across 6 of the 23 VAMCs.
- VISN E: This group consisted of 19 respondents from 5 of the 23 VAMCs.
Arm/Group | VISN A | VISN B | VISN C | VISN D | VISN E
Number analyzed (Participants) | 23 | 55 | 7 | 59 | 19
Number analyzed (VAMC) | 4 | 4 | 4 | 6 | 5
score on a scale
  Program Needs | 25.77 (7.78) | 31.74 (7.27) | 32.86 (11.47) | 28.96 (7.55) | 27.17 (10.29)
  Training Needs | 21.90 (5.25) | 25.94 (8.49) | 30.00 (13.84) | 25.93 (7.33) | 24.78 (9.64)
  Pressure for Change | 29.91 (5.04) | 30.56 (6.16) | 30.00 (6.80) | 29.29 (6.03) | 28.87 (8.74)
  Staffing | 29.86 (6.61) | 28.23 (6.64) | 30.00 (6.08) | 31.15 (6.37) | 26.67 (4.84)
  Mission | 33.46 (6.94) | 31.38 (6.96) | 32.29 (10.09) | 33.27 (6.48) | 30.21 (7.45)
  Cohesion | 31.67 (10.30) | 32.36 (8.00) | 35.24 (8.58) | 33.75 (7.56) | 33.32 (8.49)
  Autonomy | 34.78 (5.71) | 32.47 (5.75) | 32.00 (7.83) | 35.98 (4.80) | 32.24 (5.22)
  Communication | 31.74 (7.27) | 28.18 (6.87) | 29.86 (6.99) | 30.80 (7.27) | 30.32 (7.16)
  Stress | 33.19 (8.14) | 34.63 (6.93) | 30.71 (11.79) | 31.31 (8.11) | 36.97 (8.32)
  Change | 31.30 (5.74) | 29.52 (6.30) | 29.71 (11.97) | 32.72 (5.82) | 31.47 (4.63)
Statistical Analysis 1: Comparison: VISN A vs VISN B vs VISN C vs VISN D vs VISN E; Program Needs; Test type: Superiority; p = .018, ANOVA; F (4, 158) = 3.08
Statistical Analysis 2: Comparison: VISN A vs VISN B vs VISN C vs VISN D vs VISN E; Training Needs; Test type: Superiority; p = .136, ANOVA; F (4, 158) = 1.78
Statistical Analysis 3: Comparison: VISN A vs VISN B vs VISN C vs VISN D vs VISN E; Test type: Superiority — Pressure for Change; p = .812, ANOVA; F (4, 158) = 0.39
Statistical Analysis 4: Comparison: VISN A vs VISN B vs VISN C vs VISN D vs VISN E; Test type: Superiority — Staffing; p = .358, ANOVA; F (4, 158) = 1.10
Statistical Analysis 5: Comparison: VISN A vs VISN B vs VISN C vs VISN D vs VISN E; Test type: Superiority — Mission; p = .748, ANOVA; F (4, 158) = 0.48
Statistical Analysis 6: Comparison: VISN A vs VISN B vs VISN C vs VISN D vs VISN E; Cohesion; Test type: Superiority; p = .748, ANOVA; F (4, 158) = 0.48
Statistical Analysis 7: Comparison: VISN A vs VISN B vs VISN C vs VISN D vs VISN E; Autonomy; Test type: Superiority; p = .005, ANOVA; F (4, 158) = 3.88
Statistical Analysis 8: Comparison: VISN A vs VISN B vs VISN C vs VISN D vs VISN E; Communication; Test type: Superiority; p = .224, ANOVA; F (4, 158) = 1.44
Statistical Analysis 9: Comparison: VISN A vs VISN B vs VISN C vs VISN D vs VISN E; Stress; Test type: Superiority; p = .043, ANOVA; F (4, 158) = 2.52
Statistical Analysis 10: Comparison: VISN A vs VISN B vs VISN C vs VISN D vs VISN E; Change; Test type: Superiority; p = .096, ANOVA; F (4, 158) = 2.01

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious and other adverse events were not monitored or assessed for this implementation evaluation by the study team.
Description: All-cause mortality, serious and other adverse events were not monitored or assessed for this implementation evaluation by the study team.
Groups:
- VISNs Requesting Implementation Support: This cohort consists of 23 VA Medical Centers (VAMC's) needing additional implementation support to fully implement REACH VET as identified by Veteran Integrated Service Network (VISN) leadership, and that agreed to participate.
Arm/Group | VISNs Requesting Implementation Support
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT03280225/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT03280225/SAP_001.pdf